CLINICAL TRIAL: NCT06306716
Title: A Clinical Evaluation of a New NPWT Dressing
Brief Title: A Clinical Study on New Negative Pressure Wound Therapy Dressing in the Management of Chronic & Acute Wounds
Status: Terminated | Type: Observational
Why Stopped: The primary reason for this early termination is insufficient enrollment, compounded by recruitment challenges and Impending Expiry of Study Product
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LEO.2021.10
Record Dates: First submitted 2024-02-29; First posted 2024-03-12 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-09

CONDITIONS: Chronic Wounds; Acute Wounds
Keywords: Negative Pressure Wound Therapy (NPWT) Dressing; RENASYS Film with AIRLOCK Technology; Chronic and acute wounds
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Chronic and acute wounds: Subjects hospitalized due to chronic and acute wounds
  Interventions: Device: RENASYS Film with AIRLOCK Technology

INTERVENTIONS:
Device: RENASYS Film with AIRLOCK Technology — RENASYS Film with AIRLOCK Technology intended for use with Smith+Nephew RENASYS NPWT Systems
  Other Names: RENASYS Dressing

SUMMARY:
The purpose of the study is to evaluate the clinical performance of a new Negative Pressure Wound Therapy dressing in the management of chronic and acute wounds.

DETAILED DESCRIPTION:
The primary objective is to evaluate the percentage of wounds progressing to healing at the end of the treatment period. The study will also evaluate the percentage of granulation tissue, pain experienced on dressing change and safety by way of incidence and nature of device-related or procedure-related Adverse Events and Device Deficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent.
* Subject is 18 years of age or over.
* Subject is able and willing to comply with study requirements.
* Subject is suitable to participate in the study in the opinion of the Investigator. .
* Subject has a wound(s) that, per Instructions for Use (IFU), is indicated and suitable for management with NPWT and fits one of the following wound types: a. Chronic* (this may include Diabetic Foot Ulcers (DFUs), Venous Leg Ulcers (VLUs), Pressure Ulcers but this is not an exhaustive list) b. Acute (this may include traumatic and dehisced surgical wounds and partial thickness burns) *Chronic wound(s) in this study is defined as any wound of less than three months duration that is not healing after thirty (30) days of standard care and having addressed the underlying cause
* Subject's wound to be treated is of a size that can be managed with one of the available sizes of the study device

Exclusion Criteria:

* Subject has hypersensitivity to the use of the RENASYS NPWT System or its components, or a contraindication per the IFU such as: a. exposed arteries, veins, organs, or nerves b. necrotic tissue with eschar present (unless adequately debrided) c. non-enteric and unexplored fistulas d. exposed anastomotic site e. malignancy in the wound
* Subject participation in the treatment period of another clinical trial within thirty (30) days of baseline visit or during the study.
* Subject has skin features (e.g., tattoos, pre-existing scarring, etc.) which in the opinion of the investigator will interfere with the study assessments.
* For lower extremity wounds**, any subject with a wound on a limb with an inadequate arterial supply confirmed by one of the following within 14 days of treatment:

  1. Ankle Brachial Index (ABI) <0.7
  2. Toe Brachial Index (TBI) <0.5
  3. Great toe pressure <40mmHg
  4. Abnormal triphasic or biphasic waveform patterns at the ankle **This criteria is not applicable for patients having an above, or below knee amputation.
* Any subject that meets the definition of a Vulnerable Subject per ISO 14155 (i.e., individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response). Ethnic minorities will be included providing they meet other inclusion criteria.
* Subject has had the target wound for greater than three months.
* Subject has a target wound that measures <3 millimeters (mm) in maximum depth.
* Subject has untreated osteomyelitis
* Subject has active, untreated soft tissue infection.
* Subject has wounds that has been managed with NPWT in the previous four (4) weeks
* Subject has participated previously in this clinical trial.
* Subject has a history of poor compliance with medical treatment.
* Pregnancy at time of enrolment.
* Subject has a medical or physical condition that in the opinion of the Investigator would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to enroll up to 42 subjects from clinical sites in the United States and Canada with appropriate wound types including:
  * Chronic* (this may include DFUs, VLUs, Pressure Ulcers but this is not an exhaustive list)
  * Acute (this may include traumatic and dehisced surgical wounds and partial thickness burns, but this is not an exhaustive list) *Chronic wound in this study is defined as any wound of less than three months duration that is not healing after thirty (30) days of standard care and having addressed the underlying cause.
  As this is a pilot study, there are no limits to the inclusion of any particular wound type (chronic or acute) or inpatient/outpatient care at time of enrollment. Patients must be able to attend follow-up visits in clinic if they are receiving outpatient care.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Wound Healing Status | End of treatment period, up to 3 weeks
  Progression of wound healing will be assessed by the treating clinician and compared to the wound at treatment Day 0 (baseline) by recording on a 4-point Likert scale as:
  * "Wound healed"
  * "Wound progressing to healing"
  * "Wound static"
  * "Wound deteriorating"
  Any subject responding within the 2 categories of "Wound healed" or "Wound progressing to healing" will be considered a success.

SECONDARY OUTCOMES:
Percentage Reduction in Wound Volume from Baseline to Week 3 | Day 0, 1, 2, and 3 Weeks
  Percentage reduction in wound volume as measured by imaging - day 0, weekly from week 1 to week 3 of treatment or to point of wound closure if that occurs first.
Percentage Reduction in Wound Area from Baseline to Week 3 | Day 0, 1, 2, and 3 Weeks
  Percentage reduction in wound area as measured by imaging - day 0, weekly from week 1 to week 3 of treatment or to point of wound closure if that occurs first.
Percentage Reduction in Wound depth from Baseline to Week 3 | Day 0, 1, 2, and 3 Weeks
  Percentage reduction in wound depth as measured by imaging - day 0, weekly from week 1 to week 3 of treatment or to point of wound closure if that occurs first.
Percentage Area of Wound Bed Covered with Granulation Tissue | Day 0, 1, 2, and 3 Weeks
  The percentage of the wound bed covered with granulation tissue will be summarised using continuous summary statistics at day 0, weeks 1, 2 and 3 for each wound type and overall.
Peri-wound Pain Scores at Dressing Removal | Day 0, 1, 2, and 3 Weeks
  Pain scores on removal of the dressing specifically from the peri-wound skin will be assessed using a 0-100 Visual Analog Scale (VAS) scale, with zero (0) indicating no pain and 100 indicating the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Baboolal, Study Chair — Smith & Nephew, Inc.
Locations (2):
- Lawson Health Research Institute, London, Ontario, Canada
- Wound Care Plus Research and Education Center, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No